CLINICAL TRIAL: NCT00695812
Title: The Development of Younger Siblings of Children With Autism Now at 10 Years of Age
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Prof. Ruth Shalev, Shaare Zedek Medical Center, Neurology, Pediatric
Other Study IDs: Siblings Autism.ctil
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Autism Spectrum Disorders
Keywords: Neurodevelopmental disorders; Autism Spectrum Disorders; Broader autism phenotype; Siblings; Cognitive language and social emotional development; to identify siblings who manifest any autism or broader autism phenotype characteristics
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Siblings of children with Autism
- 2: Siblings of children with typical development

SUMMARY:
Background: Autism is a complex developmental disorder involving difficulties in verbal and nonverbal communication, social-emotional functioning, and markedly restricted interests and activities. Strong evidence from research conducted with family members of children with autism supports the role of genetic factors in its etiology. Thus, some family members are characterized by the broad autism phenotype (BAP) which involves a clinical picture of milder but qualitatively similar difficulties.

Working hypothesis and aims: Researchers recently initiated prospective longitudinal studies investigating the early developmental profiles of young siblings of children with autism (SIBS-A). Such longitudinal SIBS-A study is currently conducted at the Hebrew University and includes the oldest siblings studied to date. Our main aim is to identify siblings who manifest any autism or BAP characteristics.

Methods: Two groups, SIBS-A (n = 42) and siblings of children with typical development (SIBS-TD, n = 62), were seen at ages 4, 14, 24, 36, 54 months and 7 years. We plan to continue the investigation at age 10 years, a time when school related abilities and social/emotional competences are more consolidated and to investigate the developmental trajectories of children's abilities from age 4 months to 10 years using growth curve analyses.

Expected results: We expect that compared to SIBS-TD, significantly more 10-year-old SIBS-A will display difficulties related to ASD or BAP related difficulties. We also expect to identify different patterns of stability and/or change in the development of children's abilities from age 4 months to 10 years, between the two groups.

Importance: This study provides a useful approach for the examination of the main research hypothesis regarding the development of SIBS-A. One of the main advantages of using the growth curve analysis is the identification of early predictive markers for future development.

Probable implications to Medicine: This research has significant implication for early identification and the search into the causes of autism and the BAP, as well as for implementation of early treatment and prevention programs. By highlighting expressions of ASD and the BAP in siblings, we may identify early clinically predictive behavioral markers associated with their onset and contribute to the investigation of underlying genetics mechanisms.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the SIBS:

* A group comprised intact families who had a child with autism.

Inclusion criteria for families in the SIBS-TD group:

* Intact families with a newborn and an older child who exhibited typical development with no history of any learning and/or emotional difficulties according to parental report

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants in the SIBS-A and SIBS-TD groups, who are now reaching the age of 10 years, participated in the longitudinal study and were seen at the ages of 4, 14, 24, 36, 54 months and 7 years. The SIBS-A group (n = 42) comprises children who have an older sibling with autism. All probands were diagnosed using the Autism Diagnostic Observation Schedule (Lord, Rutter, DiLavore & Risi, 2002) and/or the Autism Diagnostic Interview - Revised (ADI-R; Lord, Rutter, & Le Couteur, 1994). Families were recruited through treatment centers, special schools, the national organization for children with autism in Israel, and through families of children with autism.
  The SIBS-TD group (n = 62) comprises children who have an older sibling with typical development and who participated in the longitudinal study. Families were recruited from maternity wards in Jerusalem. (more information is available in Yirmiya et al., 2006).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)